CLINICAL TRIAL: NCT00608738
Title: Developing a Nested Whole-Person-Care Guide: Screening and Evaluation Steps (American Cancer Society) ACS
Brief Title: Using Whole-Person-Care Guide in Patients Receiving Care for Cancer or Complications From Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Health Services Research
Other Study IDs: ACS 03CC1; NU-0931-005; NU-200708-1439
Record Dates: First submitted 2008-02-05; First posted 2008-02-06 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Chemotherapeutic Agent Toxicity; Infection; Malnutrition; Musculoskeletal Complications; Neutropenia; Radiation Toxicity; Thrombocytopenia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neutropenia; infection; radiation toxicity; chemotherapeutic agent toxicity; malnutrition; musculoskeletal complications; thrombocytopenia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Infections; Malnutrition; Neutropenia; Radiation Injuries; Thrombocytopenia

INTERVENTIONS:
Other: informational intervention
Other: medical chart review
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Gathering information about patients with cancer and cancer-related conditions may help doctors learn more about a patient's needs and help doctors plan the best treatment.

PURPOSE: This clinical trial is studying how well a whole-person-care guide works in identifying patient needs in patients with cancer or complications from cancer treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine what patient needs are detected from NEST13+ interviews of cancer patients and their caregivers.
* To determine the concordance among patient, caregiver, and team goals.
* To determine palliative care services provided.

OUTLINE: Participants are assigned sequentially to 1 of 2 intervention groups.

* Group 1 (NEST13+): Patients and caregivers undergo NEST13+ interviews at the time of admission to Northwestern Memorial Hospital (caregivers answer the NEST13+ interviews from the patient's perspective). A NEST13+ care plan is then derived from both patient and caregiver responses. Research MD or RN presents patient's NEST13+ findings and recommended interventions for integration with actual care. On the day of discharge, patients and caregivers undergo a second NEST13+ interview.
* Group 2 (control): Patients and caregivers undergo a sham interview at the time of admission to Northwestern Memorial Hospital. On the day of discharge, patients and caregivers undergo a NEST13+ interview as in group 1.

Medical charts for all patients are reviewed by a member of the research staff to document needs assessments in domains covered by NEST and to document palliative care-related decisions. Abstracted chart review by blinded experts is also performed to evaluate palliative care quality based on National Comprehensive Cancer Network guidelines.

PROJECTED ACCRUAL: A total of 500 patients and 250 caregivers will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of cancer
* Admitted to one of the two oncology units at Northwestern Memorial Hospital either for treatment of cancer or treatment-related complications

  * Complications include, but are not limited to, any of the following:

    * Febrile neutropenia
    * Infection
    * Esophagitis from radiochemotherapy
    * Malnutrition
    * Spinal cord compression
    * Bone pain secondary to metastatic bone disease
    * Thrombocytopenia

PATIENT CHARACTERISTICS:

* Able to read and understand English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2001-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Patient needs detected
Concordance among patient, caregiver, and team goals
Qualitative and quantitative evaluation of palliative care services provided

CONTACTS AND LOCATIONS:
Overall Officials: Linda Emanuel, MD, PhD, Study Chair — Robert H. Lurie Cancer Center